CLINICAL TRIAL: NCT03161847
Title: Natural History Study of Oculopharyngeal Muscular Dystrophy
Acronym: NH-OPMD
Status: Withdrawn | Type: Observational
Why Stopped: No subjects were enrolled
Sponsor: University of New Mexico (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 16-326
Record Dates: First submitted 2017-05-16; First posted 2017-05-22 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2017-05

CONDITIONS: Oculopharyngeal Muscular Dystrophy
Keywords: OPMD
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OPMD Subjects: The study cohort consists of individuals with genetically confirmed OPMD who will be followed longitudinally using periodic standardized assessments of clinical status in an observational, non-interventional study.
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — Non-interventional study

SUMMARY:
The objective of this study is to test a set of clinical outcome measures longitudinally in a cohort of OPMD patients to identify ones that show quantifiable change over time as the disease progresses. The investigators' goal is to delineate the natural history of OPMD.

DETAILED DESCRIPTION:
OPMD patients will undergo a screening evaluation and testing to confirm the participants carry the OPMD mutation. Subjects fulfilling the inclusion/exclusion criteria will be enrolled and followed prospectively at regular intervals to determine the natural history of this disease. Measures of muscle function and swallowing will be made at baseline and at follow-up visits to measure natural clinical progression.

ELIGIBILITY:
Inclusion Criteria:

* OPMD by genetic criteria
* ≥ 18 years old
* English-speaking

Exclusion Criteria:

* Another medical condition that precludes safe completion of study tasks (such as severe cardiac or respiratory disease)
* Another medical condition that causes symptoms similar to OPMD (i.e., ptosis, dysphagia [trouble swallowing] or limb weakness).
* History of head or neck cancer, or history of radiation to the head or neck
* A videofluoroscopic swallow study within the 12 months prior to study enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Genetically Confirmed Oculopharyngeal Muscular Dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Muscle Strength over time | Baseline and every 9 months for 3 years
  Change in Manual muscle testing over time

SECONDARY OUTCOMES:
Dysphagia severity over time | Baseline and every 9 months for 3 years
  Videofluoroscopic Swallow Studies

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Youssof, MD, MS, Principal Investigator — New Mexico Neuromuscular Center

IPD SHARING:
Plan to Share IPD: No